CLINICAL TRIAL: NCT02653170
Title: The Michigan Stroke Transitions Trial (MISTT): Improving Care Transitions for Acute Stroke Patients Through a Patient-centered Home Based Case Management Program
Brief Title: Michigan Stroke Transitions Trial
Acronym: MISTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: University of Michigan (Other); Trinity Health Michigan (Other); Sparrow Health System (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Mathew Reeves, Professor, Epidemiology, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 135457; HIS-1310-07420-01 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2015-04-09; First posted 2016-01-12 (Estimated); Results first posted 2019-08-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-07

CONDITIONS: Acute Stroke
Keywords: acute stroke; care transitions; patient engagement; patient education; caregivers; social workers
MeSH Terms: conditions — Stroke; Patient Participation | interventions — Spectinomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (No Intervention): Patients in this group will receive the hospitals' usual transitional care approach.
- SCM (Experimental): One intervention is provided:
  1. SCM (Stroke Case manager): a trained social worker who provides in-home case management services.
  Interventions: Other: SCM
- SCM and VSSP (Experimental): Two interventions are provided:
  1. SCM (Stroke Case manager): a trained social worker who provides in-home case management services. Plus:
  2. VSSP (Virtual Stroke Support Portal): Access and training in the use of the VSSP: a purpose-built, online, patient-centered information and support resource.
  Interventions: Other: SCM and VSSP

INTERVENTIONS:
Other: SCM — One intervention (SCM) is provided. Stroke Case Managers (SCMs) will conduct 2 home visits; the first within 72-96 hours and the other after 30-days of returning home. SCMs will conduct weekly follow-up phone calls. Additional home visits are permitted if needed. Home visit activities include:
  1. Biopsychosocial assessment of patient and caregiver needs.
  2. Set up appointments.
  3. Assist scheduling appointments with primary care physician and other medical providers.
  4. Promote medication adherence through medication tool kits, pill organizers and other aids.
  5. Facilitate patient and caregiver engagement and activation.
  6. Facilitate access to social and community services.
  Arms: SCM
Other: SCM and VSSP — SCM: Stroke Case Managers (SCMs) will conduct home visits at 72-96 hours and after 30-days. SCMs will conduct weekly follow-up phone calls. Additional home visits are permitted as needed. Activities include:
  1. Biopsychosocial assessment of patient and caregiver needs.
  2. Set up appointments.
  3. Assist scheduling appointments with primary care physician and other medical providers.
  4. Promote medication adherence through medication tool kits, pill organizers and other aids.
  5. Facilitate patient and caregiver engagement and activation.
  6. Facilitate access to social and community services.
  VSSP: Access and training on the Virtual Stroke Support Portal, an online information and support website which includes:
  1. Contact list of care team members.
  2. Access to hospital patient portal.
  3. Stroke education materials, resources, and guidelines.
  4. Access to Michigan 2-1-1 services.
  5. Medication information and adherence tools.
  6. Patient and Caregiver support networks.
  Arms: SCM and VSSP

SUMMARY:
The Michigan Stroke Transitions Trial (MISTT) is a patient-centered randomized control trial that aims to improve the experience of stroke patients after they return home. The MISTT study will test the effect of two complementary interventions against usual care. The two interventions include: a) Stroke Case Managers (SCMs) who are trained social workers, and b) an online informational website or portal. The 12 week intervention period begins when the stroke patient returns home from the hospital or rehab facility. The SCMs will conduct at least 2 home visits with the patient (one within 3-4 days and one around 30 days) along with weekly follow-up telephone calls. Supplemental home visits will be used as necessary over the 12 week period. At the first home visit the social workers will conduct a comprehensive in-home assessment and link patients and caregivers to local resources as necessary. Patients also assigned to the website will have access to a patient-centered online information and support resource called the Virtual Stroke Support Portal (VSSP). The investigators hypothesize that this personalized case management program will reduce patient and caregiver needs, improve quality of life, and decrease caregiver stress. The MISTT study will enroll 315 acute stroke patients discharged from 3 Michigan hospitals and will be completed by the end of 2017.

DETAILED DESCRIPTION:
To improve care transitions for acute stroke patients this pragmatic, community-based, randomized, open clinical trial will test the efficacy of two separate but complementary interventions against usual care. The parallel group design will compare the following 3 groups:

1. Usual care
2. Stroke Case Manager (SCM): trained social workers who provide home based case management services
3. SCM services plus access to the Virtual Stroke Support Portal (VSSP) an online information and support resource.

This patient-level randomized trial will be conducted at 3 Michigan hospitals and will enroll a total of 315 acute stroke patients (105 per intervention group). Each hospital will enroll cases over an 18 month period. Randomization will be balanced within each hospital to ensure that an equal number of patients are assigned to the 3 groups. If the patient identifies a primary caregivers they will be contacted and enrollment accordingly.

The trial interventions begin once the patient returns home (= Day 1) and end 3 months later (= Day 90). Outcomes data will be collected by telephone at baseline (= Day 7) and at Day 90. Subjects who are enrolled but do not go home within 1 month (because they remain in a rehabilitation or Skilled Nursing Facility) will be dropped and replaced by new patients. Two primary patient-level outcome measures include the Patient Activation Measure (PAM), a measure of self-efficacy, and the PROMIS-10, a global quality of life scale. Two primary caregiver-level outcome measures include the Bakas Caregiving Outcomes Scale (BCOS) and depression (PHQ-9).

By adhering to the principles of pragmatic trials, this trial is designed to inform typical U.S. clinical practice, with outcomes that are directly relevant to patients and caregivers. Specifically, this trial is designed to answer the practical question of whether the transitional care experience of stroke patients and caregivers can be improved by social workers who visit the home, and whether their effectiveness can be enhanced by a comprehensive patient-centered online resource.

ELIGIBILITY:
Patient Inclusion Criteria:

* A final confirmed hospital diagnosis of acute stroke (ischemic or hemorrhagic).
* Patient living at home pre-stroke.
* Presence of stroke-related deficits at admission (defined as a National Institute of Health Stroke Severity score of >=1).
* Presence of at least mild functional limitations at discharge (defined as a modified Rankin score [mRS] score of >=1), or therapy ordered.
* Discharged directly home (includes patient's residence or that of a family member).
* Discharged to a rehabilitation facility (IRF or SNF) with the expectation of return to home within 4 weeks.

Patient Exclusion Criteria:

* Patients who live more than 50 miles from the hospital (for reasons related to the home visits).
* Patients discharged to nursing home, hospice care or LTCH (Long term care hospital).
* Patients who have clinically documented cognitive deficits or stroke-related impairments including aphasia sufficient to impact the consent process and for whom a proxy respondent is not available.
* Patients who fail the 6-item cognitive screening (SIS-6) for cognitive impairment (score <=4) and for whom a proxy respondent is not available
* Patients enrolled in another acute stroke intervention trial that has a significant impact on the post-acute period (i.e., intensive data collection required of patient during follow-up).
* Limited life expectancy (< 6 months) or significant medical comorbidity likely to impact completion of the study (e.g., severe mental illness, drug or alcohol use or dependence, metastatic cancer).
* Neither the patient nor caregiver speaks English.

Caregiver Inclusion Criteria:

* Age 18 or over.
* Are identified by the stroke patient as the primary caregiver (individual who has primary responsibility for assisting with the patient's care).
* Speaks English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathew J Reeves, BVSc, PhD, Principal Investigator — Professor, Department of Epidemiology and Biostatistics, College of Human Medicine
Locations (3):
- United States (3):
  - University of Michigan, Ann Arbor, Michigan
  - Sparrow Health System, Lansing, Michigan
  - Saint Joseph Mercy Health System, Ypsilanti, Michigan

REFERENCES:
- [Background] Reeves MJ, Hughes AK, Woodward AT, Freddolino PP, Coursaris CK, Swierenga SJ, Schwamm LH, Fritz MC. Improving transitions in acute stroke patients discharged to home: the Michigan stroke transitions trial (MISTT) protocol. BMC Neurol. 2017 Jun 17;17(1):115. doi: 10.1186/s12883-017-0895-1. PMID 28623892
- [Derived] Reeves MJ, Fritz MC, Woodward AT, Hughes AK, Coursaris CK, Swierenga SJ, Nasiri M, Freddolino PP. Michigan Stroke Transitions Trial. Circ Cardiovasc Qual Outcomes. 2019 Jul;12(7):e005493. doi: 10.1161/CIRCOUTCOMES.119.005493. Epub 2019 Jul 12. PMID 31296043

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients and their caregivers were recruited from three mid-Michigan hospital stroke units. MISTT recruitment started in January 2016 and concluded in July 2017.
Pre-assignment Details: Of 320 enrolled patients, 55 were excluded prior to randomization due to extended rehab stays lasting >4 weeks (n=36), health reasons preventing participation (n=7), and other reasons that contributed to ineligibility (n=12).
  Of 210 enrolled caregivers, 41 were excluded prior to randomization due to exclusion of their patient.
Groups:
- Usual Care: Patients in this group will receive the hospitals' usual transitional care approach along with mailings of stroke and health-related brochures to help promote study retention.
- SWSCM: One intervention is provided:
  1. SWSCM (Social Work Case Management) program: a trained social worker provides in-home case management services.
  SWSCM: Stroke Case Managers (SWSCMs) will conduct 2 home visits; one within 72-96 hours and another after 30-days of returning home. SWSCMs will conduct weekly follow-up phone calls. Additional home visits are permitted as needed. Home visit activities include:
  1. Biopsychosocial assessment of patient and caregiver needs.
  2. Set up appointments.
  3. Assist scheduling appointments with primary care physician and other medical providers.
  4. Promote medication adherence through medication tool kits, pill organizers and other and activation.
  5. Facilitate patient and caregiver engagement and activation.
  6. Facilitate access to social and community services.
- SWSCM and VSSP Website: Two interventions are provided:
  1. SWSCM (Social Work Case Management) program: a trained social worker provides in-home case management services.
  2. VSSP (Virtual Stroke Support Portal): Access and training in the use of the VSSP, a purpose-built, online, patient-centered information and support resource intended to complement the SWSCM program.
  SWSCM and VSSP:
  SWSCM activities as described in the SWSCM group.
  VSSP website: Access and training on the Virtual Stroke Support Portal, an online information and support website which includes:
  1. Care team contact list
  2. Hospital patient portal access
  3. Stroke education materials and resources
  4. Access to Michigan 2-1-1 services
  5. Medication information and adherence tools
  6. Patient and Caregiver support networks
Period: Overall Study
Arm/Group | Usual Care | SWSCM | SWSCM and VSSP Website
Started (Numbers are reported for patient participants only.) | 87 | 88 | 90
Completed | 70 | 72 | 72
Not Completed | 17 | 16 | 18
Not completed — Withdrawal by Subject | 3 | 8 | 3
Not completed — withdrawn by study team | 2 | 4 | 5
Not completed — Lost to Follow-up | 12 | 4 | 10

BASELINE CHARACTERISTICS:
Groups:
- SWSCM: One intervention is provided:
  1. SWSCM (Social Work Case Management) program: a trained social worker provides in-home case management services.
  SWSCM program: Stroke Case Managers (SWSCMs) will conduct 2 home visits; one within 72-96 hours and another after 30-days of returning home. SWSCMs will conduct weekly follow-up phone calls. Additional home visits are permitted if as needed.
  1. Biopsychosocial assessment of patient and caregiver needs.
  2. Set up appointments.
  3. Assist scheduling appointments with primary care physician and other medical providers.
  4. Promote medication adherence through medication tool kits, pill organizers and other aids.
  5. Facilitate patient and caregiver engagement and activation.
  6. Facilitate access to social and community services.
- Total: Total of all reporting groups
Arm/Group | Usual Care | SWSCM | SWSCM and VSSP Website | Total
Number analyzed (Participants) | 87 | 88 | 90 | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (13.9) | 67.5 (13.0) | 66.1 (12.7) | 66.2 (13.2)
Age, Customized [Count of Participants; unit: Participants]
  Age in years: 18-54.9 | 20 | 15 | 17 | 52
  Age in years: 55-74.9 | 47 | 44 | 51 | 142
  Age in years: 75+ | 20 | 29 | 22 | 71
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 48 | 41 | 131
  Male | 45 | 40 | 49 | 134
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 66 | 68 | 75 | 209
  Race: Non-white | 21 | 20 | 15 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic | 74 | 79 | 79 | 232
Recruitment Site [Count of Participants; unit: Participants]
  Sparrow Hospital (Lansing) | 51 | 50 | 52 | 153
  St. Joseph Mercy Hospital System (Ann Arbor) | 22 | 25 | 26 | 73
  University of Michigan Health System (Ann Arbor) | 14 | 13 | 12 | 39
Required Proxy Consent [Count of Participants; unit: Participants] — Proxy consent was required if patients failed the Six-Item Cognitive Screen (score of <=4) or had clinically documented cognitive deficits or stroke-related impairments sufficient to impact the consent process:
  Participants | 8 | 13 | 12 | 33
Stroke type [Count of Participants; unit: Participants]
  Ischemic stroke | 74 | 74 | 80 | 228
  Hemorrhagic stroke | 13 | 14 | 10 | 37
Stroke Severity [Count of Participants; unit: Participants] — Stroke severity was documented at admission using the NIH-Stroke Scale (NIHSSS) or Glasgow Coma Scale (GCS). Severity was categorized as mild (NIHSS=1-5 and GCS=13-15), moderate (NIHSS=6-13 and GCS=5-12), or severe (NIHSS=14-42, GCS=3-4).
  Participants
    Mild | 66 | 60 | 64 | 190
    Moderate | 12 | 21 | 23 | 56
    Severe | 9 | 7 | 3 | 19
Modified Rankin Score (mRS) [Count of Participants; unit: Participants] — Modified Rankin Score documented at acute hospital discharge. Scores were categorized into mild (<=2) or moderate/severe (>2).
  Participants
    Mild (score <=2) | 62 | 62 | 54 | 178
    Moderate/severe (score >2) | 25 | 26 | 36 | 87
Days Between Stroke Admission and Discharge to Home [Mean (Standard Deviation); unit: days] — Duration of time from stroke admission until discharge to home. This includes acute hospital length of stay in addition to rehabilitation length of stay, if applicable.
  days | 12.4 (11.7) | 13.8 (9.7) | 14.5 (11.2) | 13.6 (10.9)
Discharge Destination [Count of Participants; unit: Participants] — Discharge destination immediately following discharge from acute stroke hospitalization.
  Participants
    Home | 49 | 32 | 36 | 117
    Inpatient Rehabilitation (IPR/IRF) | 29 | 47 | 48 | 124
    Sub-acute Rehabilitation (SAR) | 9 | 9 | 6 | 24
History of Prior Stroke [Count of Participants; unit: Participants] | 12 | 18 | 11 | 41
History of Prior Transient Ischemic Attack (TIA) [Count of Participants; unit: Participants] | 4 | 6 | 11 | 21
History of Myocardial Infarction [Count of Participants; unit: Participants] | 6 | 7 | 11 | 24
Coronary Artery Disease [Count of Participants; unit: Participants] | 17 | 16 | 25 | 58
Atrial Fibrillation [Count of Participants; unit: Participants] | 12 | 17 | 8 | 37
Diabetes [Count of Participants; unit: Participants] | 31 | 33 | 33 | 97
Hypertension [Count of Participants; unit: Participants] | 60 | 67 | 78 | 205
Hyperlipidemia [Count of Participants; unit: Participants] | 46 | 41 | 43 | 130
Living Alone Pre-Stroke [Count of Participants; unit: Participants] | 19 | 27 | 20 | 66
Caregiver consented to MISTT [Count of Participants; unit: Participants] | 58 | 57 | 54 | 169
Relationship to Consented Caregiver [Count of Participants; unit: Participants]
  spouse | 33 | 33 | 36 | 102
  Other | 25 | 24 | 18 | 67
  N/A - no caregiver consented | 29 | 31 | 36 | 96
Living with Consented Caregiver [Count of Participants; unit: Participants] | 43 | 41 | 36 | 120

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (7-days Post Discharge) to 90-days in the PROMIS-10 Global Quality of Life, Physical Health T-scores (Patient)
Description: Patient-centered questionnaire of 10 self-reported items addressing the 2 main quality-of-life domains of physical and mental health which include physical health, physical function, pain, fatigue, quality of life, mental health, satisfaction with social activities, and emotional problems. PROMIS Global-10 Physical Health Quality-of-Life is a 4-item subscale measuring general aspects of physical health using a five-point Likert scale with higher scores reflecting better quality-of-life. Raw scores are summed and converted to a T-score which has a population mean score of 50 with standard deviation of 10; higher scores indicate better QOL (0-100).
Time Frame: 7 days and 90 days post discharge
Population: Number of observations used in the analysis are larger than indicated above since both available 7-day and 90-day values were utilized (n=434)
Measure: Least Squares Mean (Standard Error); unit: change in T-score
Arm/Group | Usual Care | SWSCM | SWSCM and VSSP Website
Number analyzed (Participants) | 70 | 72 | 72
change in T-score | 0.293 (0.717) | 1.263 (0.704) | 3.663 (0.690)
Statistical Analysis 1: Comparison: Usual Care vs SWSCM vs SWSCM and VSSP Website; Data were analyzed as the change over time between treatment groups (i.e., 90-day least square mean minus 7-day least square mean) using a difference-in-differences (DID) analysis that involves a group * time interaction term; Test type: Superiority; p = 0.025, Mixed Models Analysis — P-value represents the test of the interaction term for a difference-in-differences (DID) model [i.e., 2 degree freedom test of the interaction between intervention group*time]; PROC MIXED MODEL including main effects of intervention group (UC, SWSCM, SWSCM+VSSP website) and time (7-day and 90-day) plus the interaction term; difference-in-differences (DID) p-value = 0.025 — The DID estimates contrasting the 90-day minus 7-day differences in each group are as follows: SWSCM vs Usual Care = 0.970 (p=0.335), SWSCM+VSSP vs Usual Care = 3.370 (p<0.001), SWSCM+VSSP vs SWSCM = 2.400 (p=0.016)

2. Primary Outcome: Change From Baseline (7-days Post Discharge) to 90-days in the PROMIS-10 Global Quality of Life, Mental Health T-scores (Patient)
Description: Patient-centered questionnaire of 10 self-reported items addressing the 2 main quality-of-life domains of physical and mental health which include physical health, physical function, pain, fatigue, quality of life, mental health, satisfaction with social activities, and emotional problems. PROMIS Global-10 Mental Health Quality-of-Life is a 4-item subscale measuring general aspects of physical health using a five-point Likert scale with higher scores reflecting better quality-of-life. Raw scores are summed and converted to a T-score which has a population mean score of 50 with standard deviation of 10; higher scores indicate better QOL (0-100).
Time Frame: 7 days and 90 days post discharge
Population: Number of observations used in the analysis are larger than indicated above since all available 7-day and 90-day data were utilized (n=434)
Measure: Least Squares Mean (Standard Error); unit: change in T-score
Arm/Group | Usual Care | SWSCM | SWSCM and VSSP Website
Number analyzed (Participants) | 70 | 72 | 72
change in T-score | 1.187 (0.945) | 0.123 (0.926) | 1.445 (0.907)
Statistical Analysis 1: Comparison: Usual Care vs SWSCM vs SWSCM and VSSP Website; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.562, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; difference-in-differences (DID) p-value = 0.562 — The DID estimates contrasting the 90-day minus 7-day differences in each group are as follows: SWSCM vs Usual Care = -1.064 (p=0.422), SWSCM+VSSP vs Usual Care = 0.258 (p=0.844), SWSCM+VSSP vs SWSCM = 1.322 (p=0.309)

3. Primary Outcome: Change From Baseline (7-days Post Discharge) to 90-days in the Bakas Caregiving Outcomes Scale Scores (Caregiver)
Description: Instrument designed to measure perceived caregiver life changes in response to providing care to stroke survivors. Bakas is a 15-item measure using a rating scale with 7 points ranging from -3 (changed for the worse) to +3 (changed for the best); responses are converted to a 1-7 scale and summed (range 15-105). Higher scores indicate more positive changes resulting from caregiving experience whereas lower scores indicate negative changes.
Time Frame: 7 days and 90 days post discharge
Population: Number of observations used in the analysis are larger than indicated above since all available 7-day and 90-day data were utilized (n=263)
Measure: Least Squares Mean (Standard Error); unit: change in score
Arm/Group | Usual Care | SWSCM | SWSCM and VSSP Website
Number analyzed (Participants) | 44 | 43 | 42
change in score | 1.934 (1.496) | 0.646 (1.561) | 1.961 (1.522)
Statistical Analysis 1: Comparison: Usual Care vs SWSCM vs SWSCM and VSSP Website; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.789, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline (7-days Post Discharge) to 90-days in the Patient Activation Measure Scores (Patient)
Description: Patient questionnaire to assess knowledge, skills, and self-efficacy for managing one's own healthcare. Patient Activation Measure is a 13-item survey using a five-point Likert scale (strongly disagree, disagree, agree, strongly agree, NA) whose response items are summed and converted to an activation score ranging from 0-100. Higher scores indicate a higher level of activation.
Time Frame: 7 days and 90 days post discharge
Population: Number of observations used in the analysis are larger than indicated above since all available 7-day and 90-day data were utilized (n=413)
Measure: Least Squares Mean (Standard Error); unit: change in PAM score
Arm/Group | Usual Care | SWSCM | SWSCM and VSSP Website
Number analyzed (Participants) | 70 | 72 | 72
change in PAM score | 0.874 (2.018) | -0.777 (1.958) | 5.897 (1.919)
Statistical Analysis 1: Comparison: Usual Care vs SWSCM vs SWSCM and VSSP Website; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.042, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; difference-in-differences (DID) p-value = 0.042 — The DID estimates contrasting the 90-day minus 7-day differences in each group are as follows: SWSCM vs Usual Care = -1.651 (p=0.558), SWSCM+VSSP vs Usual Care = 5.023 (p=0.073), SWSCM+VSSP vs SWSCM = 6.674 (p=0.016)

5. Secondary Outcome: Change From Baseline (7-days Post Discharge) to 90-days in Depression Symptoms (PHQ-9) (Caregiver)
Description: The Patient Health Questionnaire (PHQ-9) measures severity of depression symptoms. PHQ-9 is a 9-item measure using a four-point Likert scale (not at all, several days, more than half the days, nearly every day). Response items are summed (range 0-27) with higher scores indicating the respondent is experiencing more symptoms of depression.
Time Frame: 7 days and 90 days post discharge
Population: Number of observations used in the analysis are larger than indicated above since all available 7-day and 90-day data were utilized (n=265)
Measure: Least Squares Mean (Standard Error); unit: change in PHQ-9 score
Arm/Group | Usual Care | SWSCM | SWSCM and VSSP Website
Number analyzed (Participants) | 44 | 43 | 42
change in PHQ-9 score | -0.919 (0.537) | -1.0100 (0.560) | -0.947 (0.551)
Statistical Analysis 1: Comparison: Usual Care vs SWSCM vs SWSCM and VSSP Website; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.993, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

6. Other Pre Specified Outcome: NeuroQOL Anxiety Scale (Patient)
Description: Validated QOL scale measuring patient anxiety (administered by computer adaptive testing).
Time Frame: 90 day post discharge
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Depression Symptoms (PHQ-9) (Patient)
Description: Validated 9-item questionnaire to identify depressive symptoms.
Time Frame: 90 day post discharge
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Hospital Readmission (Patient)
Description: Unscheduled hospital admissions
Time Frame: 90 day post discharge
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Stroke Recurrence (Patient)
Description: New onset acute stroke events requiring hospital admission
Time Frame: 90 day post discharge
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Home Time (Patient)
Description: Total number of days spent at home since discharge back to home.
Time Frame: 90 day post discharge
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Oberst Caregiver Burden Scale (OCBS) (Caregiver)
Description: Validated 15-item questionnaire measuring caregiver burden in response to providing care to stroke survivors.
Time Frame: 90 day post discharge
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Unhealthy Days (Caregiver)
Description: Number of days in the past 30 days that the caregiver reported that their own physical or mental health had not been good.
Time Frame: 90-days post discharge
Reporting Status: Not Posted

13. Other Pre Specified Outcome: PROMIS Emotional Support Scale (Caregiver).
Description: A validated 4-item questionnaire measuring emotional support. Emotional support is defined as the perceived feeling of being cared for and valued as a person.
Time Frame: 90-days post discharge
Reporting Status: Not Posted

14. Other Pre Specified Outcome: PROMIS Informational Support Scale (Caregiver).
Description: A validated 4-item questionnaire measuring informational support. Informational support is defined as the perceived availability of helpful information or advice.
Time Frame: 90-days post discharge
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 90-day study participation period
Description: Serious Adverse Event: reported if admitted to Hospice Care or a Nursing Home/Long-term Care Facility Other Adverse Event: not collected
  NOTE: hospital readmissions were collected as a secondary outcome measure and were not included in the Adverse Event reporting.
Arm/Group | Usual Care | SWSCM | SWSCM and VSSP Website
All-Cause Mortality (participants affected / at risk) | 0/87 | 2/88 | 0/90
Serious Adverse Events (participants affected / at risk) | 1/87 | 2/88 | 5/90
Other Adverse Events (participants affected / at risk) | 0/87 | 0/88 | 0/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=87) | SWSCM (N=88) | SWSCM and VSSP Website (N=90)
Admitted to Nursing Home or Long-term Care Facility (General disorders) | 0 (0) | 1 (1) | 3 (3) — Admitted to nursing home or long-term care facility
Admitted to Hospice Care (General disorders) | 1 (1) | 1 (1) | 2 (2) — Admitted to Hospice Care

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-08-19): https://cdn.clinicaltrials.gov/large-docs/70/NCT02653170/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT02653170/SAP_001.pdf